CLINICAL TRIAL: NCT02412657
Title: Impact of Two Doses of Intravenous Dexamethasone on the Analgesic Duration of a Single-shot Interscalene Block With Ropivacaine for Shoulder Arthroscopy; a Prospective, Randomized, Placebo-controlled Study
Brief Title: Intravenous Dexamethasone to Increase the Analgesic Duration of Interscalene Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Veronique Brulotte, Dre Veronique Brulotte, MD, M.Sc, FRCPC, anesthesiologist, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: dexaISB
Record Dates: First submitted 2015-03-12; First posted 2015-04-09 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Dexamethasone; Calcium Dobesilate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dexamethasone 10 mg intravenous (Experimental): Dexamethasone 10 mg diluted with Normal Saline 17,5 mL i.v. (20 mL total) injected slowly during 30 seconds immediately after performing interscalene brachial plexus block
  Interventions: Drug: Dexamethasone
- Dexamethasone 4 mg intravenous (Experimental): Dexamethasone 4 mg diluted with Normal Saline 19 mL i.v. (20 mL total) injected slowly during 30 seconds, immediately after performing interscalene brachial plexus block
  Interventions: Drug: Dexamethasone
- Normal Saline 20 mL intravenous (Placebo Comparator): Normal saline 20 mL injected slowly during 30 seconds, immediately after performing interscalene brachial plexus block
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexamethasone — After the performance of inter scalene plexus blockade, patients will either receive dexamethasone 10 mg i.v. (diluted with 17.5 mL normal saline), dexamethasone 4 mg i.v. (diluted with 19 mL normal saline), or normal saline 20 ml i.v.
  Other Names: decadron
  Arms: Dexamethasone 10 mg intravenous; Dexamethasone 4 mg intravenous
Drug: Normal Saline
  Arms: Normal Saline 20 mL intravenous

SUMMARY:
Interscalene brachial plexus block provides excellent but time limited analgesia. Intravenous dexamethasone increases the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder arthroscopic surgery. We want to evaluate the effect of two different doses (dexamethasone 10 mg i.v. vs 4 mg i.v. vs placebo) on the analgesic duration of a single-shot inter scalene block. Our study hypothesis is that dexamethasone 4 mg i.v. is equivalent to dexamethasone10 mg i.v. in prolonging the analgesic duration of a single-shot interscalene block with ropivacaine.

DETAILED DESCRIPTION:
75 patients will be randomly assigned to three groups:

* D10: dexamethasone 10 mg I.V. diluted in normal saline 20cc, immediately after inter scalene block
* D4: dexamethasone 4 mg I.V. diluted in normal saline 20cc, immediately after inter scalene block
* C: control: Normal saline 20cc I.V., immediately after inter scalene block. These patient will be recruited from 3 hospitals, with two surgeons performing the surgeries.

All patients will have their surgery under regional anesthesia only provided by the inter scalene plexus block, with ropivacaine 0.5% 20cc.

In the postoperative period, patients will be given analgesic medication on an as needed basis. They will be instructed to take the first analgesic medication once postoperative shoulder pain has reached >3/10. They will note the time and day at which this outcome occurs.

ELIGIBILITY:
Inclusion Criteria:

* Elective shoulder arthroscopy under ropivacaine single-shot interscalene brachial plexus block anesthesia (rotator cuff repair and shoulder decompression)
* ASA I-III
* Age 18-80 years old

Exclusion Criteria:

* Any contraindication to interscalene brachial plexus block anesthesia
* Interscalene brachial plexus block failure
* Known local anesthetics allergy
* Dexamethasone allergy or intolerance
* Any contraindication to acetaminophen
* Any contraindication to morphine or hydromorphone
* Brachial plexus neuropathies
* Chronic pain syndrome other than shoulder pain
* Routine use of opioid medication
* Routine use of systemic corticosteroid
* Pregnancy
* Weight below 50 kilograms
* Incapability to understand a numeric verbal pain scale
* Incapability to consent
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Brulotte, MD MSc FRCPC, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (3):
- Canada (3):
  - Hopital Pierre-Boucher, Longueuil, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hopital Hotel-Dieu de Sorel, Sorel-Tracy, Quebec

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chalifoux F, Colin F, St-Pierre P, Godin N, Brulotte V. Low dose intravenous dexamethasone (4 mg and 10 mg) significantly prolongs the analgesic duration of single-shot interscalene block after arthroscopic shoulder surgery: a prospective randomized placebo-controlled study. Can J Anaesth. 2017 Mar;64(3):280-289. doi: 10.1007/s12630-016-0796-6. Epub 2017 Jan 3. PMID 28050801

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Saline 20 mL Intravenous: Normal saline 20 mL injected slowly during 30 seconds, immediately after performing interscalene brachial plexus block
  Normal Saline
Period: Overall Study
Arm/Group | Dexamethasone 10 mg Intravenous | Dexamethasone 4 mg Intravenous | Normal Saline 20 mL Intravenous
Started | 25 | 25 | 25
Completed | 24 | 23 | 22
Not Completed | 1 | 2 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone 10 mg Intravenous | Dexamethasone 4 mg Intravenous | Normal Saline 20 mL Intravenous | Total
Number analyzed (Participants) | 24 | 23 | 22 | 69
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 49 [44 to 54] | 54 [50 to 59] | 55 [51 to 58] | 53 [33 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 11 | 29
  Male | 17 | 12 | 11 | 40
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 23 | 22 | 69

OUTCOME MEASURES:

1. Primary Outcome: Duration of Analgesia
Description: Defined as the time between the performance of the block and the first analgesic request
Time Frame: 48 hours after surgery
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Dexamethasone 10 mg Intravenous | Dexamethasone 4 mg Intravenous | Normal Saline 20 mL Intravenous
Number analyzed (Participants) | 24 | 23 | 22
hours | 19.1 [11.5 to 22.8] | 19.6 [16 to 22.2] | 11.8 [8.7 to 13.8]

2. Secondary Outcome: Pain Scores
Description: On a 11-points Verbal Numeric Scale 0-10 (0= no pain, 10= worst conceivable pain)
Time Frame: every 6 hours during the first 48 hours after surgery
Reporting Status: Not Posted

3. Secondary Outcome: Residual Motor Block
Description: Scale of 0-2 (0:inability to move fingers, 1: fingers able to move, with diminished strength compared to non operated side, 2: No motor weakness of the fingers)
Time Frame: 24 hours and 48 hours
Reporting Status: Not Posted

4. Secondary Outcome: Sleep Disturbance
Description: Sleep disturbance scale 0-10 (0: no sleep disturbance from pain, 10: worst conceivable sleep disruption from pain)
Time Frame: 24 hours and 48 hours
Reporting Status: Not Posted

5. Secondary Outcome: Patients Overall Satisfaction
Description: categorical data (1: very satisfied, would recommend this analgesia protocol to others, 0: not satisfied, would not recommend this analgesia protocol to others
Time Frame: 48 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Dexamethasone 10 mg Intravenous | Dexamethasone 4 mg Intravenous | Normal Saline 20 mL Intravenous
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No